CLINICAL TRIAL: NCT05530135
Title: Life-Style Interventions for Modulating the Brain Phenotype of Takotsubo Cardiomyopathy - the BREAKOUT Study
Brief Title: Life-style Interventions for Modulating the Brain Phenotype of Takotsubo Cardiomyopathy
Acronym: BREAKOUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 283639
Record Dates: First submitted 2022-08-30; First posted 2022-09-07 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Takotsubo Cardiomyopathy
Keywords: Takotsubo Cardiomyopathy
MeSH Terms: conditions — Takotsubo Cardiomyopathy | interventions — Resistance Training; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Three arm pilot feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Placebo Comparator): Takotsubo patients receiving standard care
  Interventions: Other: Standard clinical care
- Exercise Group (Active Comparator): Takotsubo patients who will undergo an exercise program in addition to standard care
  Interventions: Other: Exercise program; Other: Standard clinical care
- CBT Group (Active Comparator): Takotsubo patients who will receive cognitive behavioural therapy in addition to standard care
  Interventions: Other: Cognitive behavioural therapy; Other: Standard clinical care

INTERVENTIONS:
Other: Exercise program — Exercise program
  Arms: Exercise Group
Other: Cognitive behavioural therapy — Cognitive behavioural therapy
  Arms: CBT Group
Other: Standard clinical care — Standard clinical care

SUMMARY:
Takotsubo cardiomyopathy presents like a heart attack and is typically triggered by intense emotional or physical stress. Recovery of this condition varies and many patients continue to suffer from symptoms such as fatigue and breathlessness for a protracted period after their event. The purpose of this study is to establish whether following a structured exercise program or a mental wellbeing program compared to usual care for 12 weeks after an episode of Takotsubo will result in significant improvement in the brain activity, general and mental wellbeing of patients.

DETAILED DESCRIPTION:
Takotsubo cardiomyopathy is characterised by sudden onset left ventricular dysfunction precipitated by major stress. This neuro-cardiac condition has a 5-year morbidity and mortality comparable with acute myocardial infarction and no current therapies exist. The psycho-somatic basis of Takotsubo suggests that its neuro-biology could be amenable to modulation. Here, the investigators propose a mechanistic three-arm pilot feasibility trial of standardised physical exercise training, cognitive behavioural therapy and current standard of care in patients who suffered a very recent episode of takotsubo cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with takotsubo cardiomyopathy in the previous three weeks
* Participant who is willing and able to give informed consent for participation in the study.
* Participant who is willing to travel to Aberdeen Royal Infirmary for the study visits.
* Healthy volunteers (for blood and saliva samples only) willing to give informed consent for participation in the study. Healthy volunteers should not be on any medication.
* For influenza T-Cell testing: healthy volunteers who have recently received their annual flu vaccination.
* Myocardial Infarction (MI) comparators: patients with type 1 acute MI (diagnosed within the last three weeks)

Exclusion Criteria:

* Any patient whose takotsubo cardiomyopathy was triggered by a physical illness that would preclude them from taking part in a physical exercise training program
* Any patient who is not able or willing to travel to the cardiovascular research facility for their study visits
* Any patient who is not able to commit to a 12 week supervised training program
* Inability to exercise on a cycle ergometer or a treadmill (e.g. use of walking aids or prosthetic limbs or advanced frailty)
* Unwillingness to participate
* Contraindication to MRI scanning such as implantable cardiac devices.
* Pregnancy
* Healthy volunteers taking medication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Hippocampal volume change | At ≤3 weeks of diagnosis of takotsubo cardiomyopathy and repeated at completion of 12 weeks intervention
  Brain Magnetic Resonance Imaging

SECONDARY OUTCOMES:
Mental wellbeing testing | At ≤3 weeks of diagnosis of takotsubo cardiomyopathy and repeated at completion of 12 weeks intervention
  Eysenck personality questionnaires, Hospital Anxiety and Depression, Perceived Stress Scale and Work & Social Adjustment
Mental wellbeing testing | At ≤3 weeks of diagnosis of takotsubo cardiomyopathy and repeated at completion of 12 weeks intervention
  Blood will be collected for PBMCs isolation and serum cytokine levels
Mental wellbeing test | At ≤3 weeks of diagnosis of takotsubo cardiomyopathy and repeated at completion of 12 weeks intervention
  Cortisol Awakening Response
Exercise Capacity | At ≤3 weeks of diagnosis of takotsubo cardiomyopathy and repeated at completion of 12 weeks intervention
  6 minute walk test and Cardiopulmonary Exercise Test
Cardiac Imaging | At ≤3 weeks of diagnosis of takotsubo cardiomyopathy and repeated at completion of 12 weeks intervention
  Echocardiography

CONTACTS AND LOCATIONS:
Locations (1):
- Aberdeen Royal Infirmary, Aberdeen, Scotland, United Kingdom